CLINICAL TRIAL: NCT03276676
Title: [18F]Fluciclovine and [18F]FLT PET/CT Assessment of Primary High-Grade Brain Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: poor accrual and PI retired
Sponsor: University of Utah (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCI104704
Record Dates: First submitted 2017-09-05; First posted 2017-09-08 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-10

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — alovudine; fluciclovine F-18

STUDY DESIGN:
Intervention Model Description: Both arms will undergo the same interventions, however, Group A will undergo three imaging sessions and Group B will undergo one imaging session
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Participants enrolled in Group A will undergo a maximum of 6 scans throughout this study. [18F]FLT- and [18F]Fluciclovine-PET/CT scans at up to three imaging time points: (1) prior to any tumor-directed therapy, (2) within 1-4 weeks after the conclusion of the intitial (~6-8 weeks) chemoradiotherapy, and (3) following suspected recurrence/progression versus treatment effect (pseudoprogression) shown with MRI, within 6 months of the completion of chemoradiation
  Interventions: Drug: [18F]FLT; Drug: [18F]Fluciclovine
- Group B (Experimental): Participants enrolled in Group B will undergo 2 scans as part of this study. [18F]FLT- and [18F]Fluciclovine-PET/CT scans will be acquired at a single timepoint, at the time of suspected pseudoprogression.
  Interventions: Drug: [18F]FLT; Drug: [18F]Fluciclovine

INTERVENTIONS:
Drug: [18F]FLT — PET exams of [18F]FLT will be acquired in each patient at up to three time points: (1) prior to any tumor-directed therapy, either prior to surgery or immediately after surgery providing a complete surgical resection was not performed and confirmed by a post-operative contrast MRI scan where residual tumor > 1.0 cm in diameter was present and prior to any tumor-directed therapy; (2) at the conclusions of the initial (~6-8 weeks) chemoradiotherapy; and (3) patients with MRI-documented possible recurrence/progression versus treatment effect (pseudoprogression) within 6 months from the time of completion of chemoradiation.
Drug: [18F]Fluciclovine — PET exams of [18F]Fluciclovine will be acquired in each patient at up to three time points: (1) prior to any tumor-directed therapy, either prior to surgery or immediately after surgery providing a complete surgical resection was not performed and confirmed by a post-operative contrast MRI scan where residual tumor > 1.0 cm in diameter was present and prior to any tumor-directed therapy; (2) at the conclusions of the initial (~6-8 weeks) chemoradiotherapy; and (3) patients with MRI-documented possible recurrence/progression versus treatment effect (pseudoprogression) within 6 months from the time of completion of chemoradiation.

SUMMARY:
The hypothesis of this exploratory clinical trial in patients with high-grade a primary brain tumor who receive chemoradiation is that the PET imaging agents [18F]Fluciclovine and/or [18F]FLT will be a better predictor of tumor response than standard MRI based brain tumor response criteria. When used in conjunction, the two PET agents may be better able to predict tumor aggressiveness and thus overall survival than the use of individual-tracer PET biomarkers. This may eventually lead to improved assessment of response (including time to progression and overall survival) and differentiation of tumor recurrence/progression from treatment effect (pseudoprogression).

DETAILED DESCRIPTION:
The standard treatment approach for patients with high-grade primary brain tumors includes maximum feasible surgical resection, followed by 6 weeks of concurrent cranial irradiation, and daily low-dose temozolomide chemotherapy; followed by 12 cycles of high-dose temozolomide administered for 5 consecutive days every 4 weeks (Stupp et al., 2005). Contrast-enhanced MRI is the current standard for evaluating the success of therapy and monitoring for tumor recurrence. MRI is typically obtained prior to initial surgery, within 24 hours after surgery, at the conclusions of cranial irradiation, and then every 8 weeks during temozolomide chemotherapy until evidence of recurrence. Despite this careful clinical and radiographic surveillance, and despite decades of research into the histologic and molecular classification of primary brain tumors, our ability to predict tumor behavior remains very limited. Some gliomas will result in overall survival times of only months, whereas other histologically-identical gliomas may yield survivals of years to decades (Curran et al., 1993, Carson et al., 2007). Current assessment of tumor response to therapy is also poor. Patients with complete radiographic response after cranial irradiation often progress rapidly post-irradiation. In contrast, some patients with enhancing masses at the end of chemoradiotherapy may respond dramatically to further chemotherapy alone; or the masses may even disappear in the absence of further therapy, so called "tumor pseudoprogression" (Chamberlain et al., 2007). This confounding situation demonstrates a need for better assessment of tumor response.

Improvements in the ability to predict tumor behavior prior to the start of therapy would allow more efficient and effective tumor surveillance; better prognostication; and more appropriate assignment of patients to conventional, aggressive, or investigational therapies early in their clinical courses. This would provide huge economic and social benefits, and could afford decisive insights into brain tumor physiology and biology.

Similarly, the ability to identify, earlier and more accurately, whether individual patients were responding to therapy would allow prompt discontinuation of ineffectual treatments and institution of potentially more effective therapies.

Previous efforts using imaging for such tasks have generally been limited to a single modality (e.g. MRI) and/or single-tracer (e.g. FDG-PET). However, there is a significant and growing body of evidence that complementary imaging of multiple aspects of tumor physiology (i.e. using multiple PET tracers) can provide greatly enhanced information over imaging with a single modality or tracer alone. In solid tumors, complex interactions exist between blood flow, metabolic activity, and oxygen status which affect metastatic and proliferative activity. Heterogeneous tumors may contain both slow-growing and fast-growing regions that present different profiles of proliferation rates and amino acid uptake.

ELIGIBILITY:
Inclusion Criteria:

* Two adult patient groups will be eligible for inclusion in this study:

Group A: Patients where there is compelling evidence, based on the MRI and/or CT imaging, that a high-grade primary brain tumor is present. Pathologic confirmation will occur with biopsy or surgery.

Patients whose tumor is felt to be inoperable and a biopsy is performed but no surgery.

Patients with a newly diagnosed primary malignant brain tumor (WHO Grade III or IV) who will be receiving chemoradiation and who either did not undergo surgical resection or underwent incomplete resection with residual tumor > 1.0 cm in greatest diameter by contrast MRI postoperatively.

Group B: Patients with pathologically proven malignant brain tumor (WHO Grade III or IV glial-based tumors) who have undergone chemoradiation and have MRI-documented possible recurrence/progression versus treatment effect (pseudoprogression) within 6 months from the time of completion of chemoradiation.

* Patients must be 18 years or older for inclusion in this study. There is little experience with the safety of [18F]FLT or [18F]Fluciclovine in children, and the risks associated with radiation exposure may be increased for children under 18 years old as well.
* Patients must document their willingness to be followed for at least 24 months after recruitment by signing informed consent documenting their agreement to have clinical endpoints and the results of histopathologic tissue analysis (when tissue becomes available from routine care) entered into a research database.
* All patients, or their legal guardians, must sign a written informed consent and HIPAA authorization in accordance with institutional guidelines.
* Determination of pregnancy status: Female patients who are not postmenopausal or surgically sterile will undergo a serum pregnancy test prior to each set of [18F]FLT and [18F]Fluciclovine PET scans. A negative test will be necessary for such patients to undergo research PET imaging.
* Pre-imaging laboratory tests must be performed within 28 days prior to the [18F]FLT imaging procedure. These must be less than 4.0 times below or above the upper or lower limit range for the respective laboratory test for entry into the study (unless clinically not relevant). In those instances where a laboratory value is outside of this range, then such a patient will be ineligible for enrollment unless at the discretion of the PI the abnormal lab value is of no clinical significance to the safety or integrity of the study results. . For follow-up scanning sessions after therapy has been instituted, laboratory testing will also be required due to the use of [18F]FLT. The patients have brain tumors and will have received chemoradiation; therefore, many routine laboratory tests may not be within the typical normal range. As such, a factor of 4.0 times above or below the upper or lower value for the normal range for any laboratory test will also be used to determine the acceptable range for the 2nd and possibly 3rd imaging time points (unless clinically not relevant as explained above). The baseline laboratory testing will include liver enzymes (ALT, AST), bilirubin (total), serum electrolytes, CBC with platelets, prothrombin time, partial thromboplastin time, BUN, and creatinine. For those patients receiving coumadin or another anticoagulant the upper limit for prothrombin time or partial thromboplastin time must not exceed 6 times the upper limit of the normal range. (Appendix E, Laboratory Study Results).

Exclusion Criteria:

* Patients with clinically significant signs of uncal herniation, such as acute pupillary enlargement, rapidly developing motor changes (over hours), or rapidly decreasing level of consciousness, are not eligible.
* Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals. Patients with significant drug or other allergies or autoimmune diseases may be enrolled at the Investigator's discretion.
* Patients who are pregnant or lactating or who suspect they might be pregnant. Serum pregnancy tests will be obtained prior to each set of multi-tracer PET scans in female patients that are not postmenopausal or surgically sterile.
* Adult patients who require monitored anesthesia for PET scanning.
* Patients who are too claustrophobic to undergo PET scanning.
* Known HIV positive patients due to the previous toxicity noted with [18F]FLT in this patient group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2023-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Yap, PhD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Group A will consist of patients from three different eligibility cohorts. The first, for patients where there is compelling evidence, based on the MRI and/or CT imaging, that a high-grade primary brain tumor is present. Pathologic confirmation will occur with subsequent biopsy or surgery. The second cohort of patients are individuals where the tumor is felt to be inoperable and a biopsy is performed but no surgery. The third cohort of patients are post-surgery where a complete surgical resection was not possible. This will be confirmed by a post-operative contrast MRI/CT scan where residual tumor > 1.0 cm in diameter is present.
  Participants enrolled in Group A will undergo a maximum of 6 scans throughout this study. [18F]FLT- and [18F]Fluciclovine-PET/CT scans at up to three imaging time points: (1) prior to any tumor-directed therapy, (2) within 1-4 weeks after the conclusion of the intitial (~6-8 weeks) chemoradiotherapy, and (3) following suspected recurrence/progression versus treatment effect (pseudoprogression) shown with MRI, within 6 months of the completion of chemoradiation.
- Arm B: Group B will enroll patients with pathologically proven malignant brain tumor (WHO Grade III or IV glialbased tumors) who have undergone chemoradiation and have a contrast enhancing mass ≥ 1.0 cm in greatest diameter concerning for pseudoprogression if MRI-documented possibility of recurrence/progression versus treatment effect (pseudoprogression) is within 6 months from the time of completion of chemoradiation.
  Participants enrolled in Group B will undergo 2 scans as part of this study. [18F]FLT- and [18F]Fluciclovine-PET/CT scans will be acquired at a single timepoint, at the time of suspected pseudoprogression.
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 4 | 6
Completed | 2 | 5
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group A: Group A will consist of patients from three different eligibility cohorts. The first, for patients where there is compelling evidence, based on the MRI and/or CT imaging, that a high-grade primary brain tumor is present. Pathologic confirmation will occur with subsequent biopsy or surgery. The second cohort of patients are individuals where the tumor is felt to be inoperable and a biopsy is performed but no surgery. The third cohort of patients are post-surgery where a complete surgical resection was not possible. This will be confirmed by a post-operative contrast MRI/CT scan where residual tumor > 1.0 cm in diameter is present.
  Participants enrolled in Group A will undergo a maximum of 6 scans throughout this study. [18F]FLT- and [18F]Fluciclovine-PET/CT scans at up to three imaging time points: (1) prior to any tumor-directed therapy, (2) within 1-4 weeks after the conclusion of the intitial (~6-8 weeks) chemoradiotherapy, and (3) following suspected recurrence/progression versus treatment effect (pseudoprogression) shown with MRI, within 6 months of the completion of chemoradiation.
- Group B: Group B will enroll patients with pathologically proven malignant brain tumor (WHO Grade III or IV glialbased tumors) who have undergone chemoradiation and have a contrast enhancing mass ≥ 1.0 cm in greatest diameter concerning for pseudoprogression if MRI-documented possibility of recurrence/progression versus treatment effect (pseudoprogression) is within 6 months from the time of completion of chemoradiation.
  Participants enrolled in Group B will undergo 2 scans as part of this study. [18F]FLT- and [18F]Fluciclovine-PET/CT scans will be acquired at a single timepoint, at the time of suspected pseudoprogression.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.87 (16.64) | 54.46 (17.93) | 49.82 (17.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Count of Patients Showing >25% Reduction in Cerebral Uptake of [18F]FLT and [18F]Fluciclovine
Description: Cerebral uptake of [18F]FLT and [18F]Fluciclovine measured in terms of SUVmax and SUVmean at each imaging time point ((1) prior to any tumor-directed therapy, (2) within 1-4 weeks after the conclusion of the initial (~6-8 weeks) chemoradiotherapy, and (3) following suspected recurrence/progression versus treatment effect (pseudoprogression) shown with MRI, within 6 months of the completion of chemoradiation). Using the first time point as baseline for the following two time points, the percent change is calculated from SUVmean and SUVmax for each of the radiotracers studied in this trial.
  This measure only applies to Group A, as multiple time points of scan data are needed to calculate change in uptake.
Time Frame: (1) Baseline [18F]FLT and [18F]Fluciclovine scans were acquired prior to initiating therapy, follow-up scans were acquired (2) 1-4 weeks following conclusion of initial chemoradiation, and (3) within 6 months of completion of chemoradiation.
Population: Only two participants from Group A were evaluable for this outcome. This outcome measure is not applicable to Group B.
Measure: Count of Participants; unit: Participants
Groups:
- Group A: Participants enrolled in Group A had a maximum of 6 scans throughout this study. [18F]FLT- and [18F]Fluciclovine-PET/CT scans at up to three imaging time points:
  1. prior to any tumor-directed therapy,
  2. within 1-4 weeks after the conclusion of the intitial (~6-8 weeks) chemoradiotherapy, and
  3. following suspected recurrence/progression versus treatment effect (pseudoprogression) shown with MRI, within 6 months of the completion of chemoradiation
Arm/Group | Group A
Number analyzed (Participants) | 2
Participants
  SUVmean (FLT) - Time Point 2: >25% Reduction | 1
  SUVmean (FLT) - Time Point 2: <=25% Reduction | 1
  SUVmax (FLT) - Time Point 2: >25% Reduction | 1
  SUVmax (FLT) - Time Point 2: <=25% Reduction | 1
  SUVmean (FLT) - Time point 3: >25% Reduction | 1
  SUVmean (FLT) - Time point 3: <=25% Reduction | 1
  SUVmax (FLT) - Time Point 3: >25% Reduction | 0
  SUVmax (FLT) - Time Point 3: <=25% Reduction | 2
  SUVmean (Fluciclovine) - Time Point 3: >25% Reduction | 1
  SUVmean (Fluciclovine) - Time Point 3: <=25% Reduction | 1
  SUVmax (Fluciclovine) - Time point 2: >25% Reduction | 1
  SUVmax (Fluciclovine) - Time point 2: <=25% Reduction | 1
  SUVmean (Fluciclovine) - Time Point 2: >25% Reduction | 1
  SUVmean (Fluciclovine) - Time Point 2: <=25% Reduction | 1
  SUVmax (Fluciclovine) - Time Point 3: >25% Reduction | 1
  SUVmax (Fluciclovine) - Time Point 3: <=25% Reduction | 1

ADVERSE EVENTS:
Time Frame: Adverse event assessment occurs through the administration of the [18F]FLT- and [18F]Fluciclovine administrations and questioned following the conclusion of the PET/CT scans. Survival was assessed until study closure, or for up to 4 years, 10 months, and 26 days after the start of the study intervention.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 4/4 | 4/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 3/4 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=4) | Group B (N=6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headach (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT03276676/Prot_SAP_002.pdf